CLINICAL TRIAL: NCT01450904
Title: The Recovery Time of Quadriceps Strength After Total Knee Arthroplasty: The Effect of Quadriceps Incision Length
Brief Title: The Recovery Time of Quadriceps Strength After Total Knee Arthroplasty (TKA): The Effect of Quadriceps Incision Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si051/2554(EC2)
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): The length of Quadriceps incision was less than 2 cm.
  Interventions: Procedure: Quadriceps incision < 2 cm
- Group B (Experimental): The length of Quadriceps incision was 2 to 4 cm.
  Interventions: Procedure: Quadriceps incision 2-4 cm
- Group C (Experimental): The length of Quadriceps incision was more than 4 cm.
  Interventions: Procedure: Quadriceps incision > 4 cm

INTERVENTIONS:
Procedure: Quadriceps incision < 2 cm — MIS-TKA was performed with less than 2 cm Quadriceps incision length
  Arms: Group A
Procedure: Quadriceps incision 2-4 cm — MIS-TKA was performed with 2 to 4 cm Quadriceps incision length
  Arms: Group B
Procedure: Quadriceps incision > 4 cm — MIS-TKA was performed with more than 4 cm Quadriceps incision length
  Arms: Group C

SUMMARY:
Minimally invasive total knee arthroplasty (MIS-TKA) became the popular technique. It had the less postoperative pain and shorter recovery time compared to the conventional technique. With using MIS technique, less cut of quadriceps tendon was the key. It related to keep more quadriceps strength and improve functional performance after TKA. However, there was no previous studies about the effect of quadriceps incision length in the recovery time of the quadriceps strength. The investigators hypothesized that longer quadriceps incision affected the longer recovery time of quadriceps strength in MIS-TKA.

ELIGIBILITY:
Inclusion Criteria:

* The patients who diagnosed primary osteoarthritis of knee with

  1. varus or valgus deformity < 20 degrees
  2. preoperative range of motion > 90 degrees
  3. extension lag < 10 degrees
  4. Flexion contracture < 30 degrees

Exclusion Criteria:

* Bilateral simultaneous total knee arthroplasty
* Previous knee surgery
* Inadequate exposure during the surgery

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The recovery time of Quadriceps strength | Upto 6 months
  Quadriceps strength was tested every month postoperatively, Recovery time was the amount of months which the Quadriceps strength returned to preoperative level.

CONTACTS AND LOCATIONS:
Overall Officials: Keerati Charoencholvanich, MD, Principal Investigator — Mahidol University